CLINICAL TRIAL: NCT04489082
Title: Use of Near Infrared Laser Stimulation for Treatment of Depression, Anxiety, Neurodegenerative Conditions, and Traumatic Brain Injury/Chronic Traumatic Encephalopathy
Brief Title: Near-Infrared Laser Stimulation for Various Neurological Conditions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20192916
Record Dates: First submitted 2020-07-21; First posted 2020-07-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Refractory Depression; Anxiety Disorders; Neurodegenerative Diseases; Traumatic Brain Injury; Chronic Traumatic Encephalopathy
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Anxiety Disorders; Neurodegenerative Diseases; Brain Injuries, Traumatic; Chronic Traumatic Encephalopathy

STUDY DESIGN:
Intervention Model Description: The present study is being undertaken as an open-label study to evaluate the safety and feasibility of near infrared therapy as an intervention for patients with refractory depression, anxiety, cognitive impairment due to a neurodegenerative disease (e.g., Alzheimer's), and traumatic brain injury.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Near Infrared Laser Therapy (Experimental): On the days of each near-infrared therapy session, patients will undergo 10 minutes of transcranial infrared laser stimulation.
  The laser dose for all conditions will be a 3.4 W continuous laser wave, at a 1064 wavelength, with irradiance (power density) at 250 milli-Watts/cm2. All groups will have treatment once a week (10 minutes per session) for 5-6 weeks. For Alzheimer's, the site targeted will be the right prefrontal cortex. Parkinson's patients will have laser delivered to the brain stem, bilateral temporal lobes. TBI/CTE patients will have the laser stimulation site dependent on location of injury. Patients with depression/anxiety will have laser stimulation applied to the prefrontal area of the head.
  Interventions: Device: Near Infrared Laser Stimulation

INTERVENTIONS:
Device: Near Infrared Laser Stimulation — 10 minutes of transcranial near infrared laser stimulation

SUMMARY:
The study will evaluate the safety and feasibility of near infrared therapy as an intervention for patients with refractory depression, anxiety, neurodegenerative disease, and traumatic brain injury.

DETAILED DESCRIPTION:
The present study is being undertaken as an open-label study to evaluate the safety and feasibility of near infrared therapy as an intervention for patients with refractory depression, anxiety, cognitive impairment due to a neurodegenerative disease (e.g., Alzheimer's), and traumatic brain injury. Baseline and outcome measures in this study utilize validated tests that are appropriate for repeated measures. The present study can be easily implemented because instruments have been in routine clinical deployment providing for a high degree of availability and reliability. Quality assurance is tightly controlled. The study population is sufficiently broad and the conditions of interest are sufficiently prevalent so that recruitment of subjects is not a limiting factor.

ELIGIBILITY:
Inclusion Criteria (depression):

* Diagnosis of Major Depressive Disorder
* Score greater than 13 on the Beck Depression Inventory
* Failure to remit with 3 antidepressants
* At least 18 years of age

Inclusion Criteria (anxiety):

* Diagnosis of Generalized or Acute Anxiety Disorder
* Score greater than 22 on the Beck Anxiety Inventory
* Failure to remit with 3 anxiolytics
* At least 18 years of age

Inclusion Criteria (neurodegenerative dementia):

* Cognitive decline with mild cognitive impairment (Clinical Dementia Rating stage 0.5) through moderate dementia (CDR stage 2)
* Lumbar puncture for Abeta 42 and Tau proteins evincing clinical correlation of neurodegenerative disease pathology
* Advanced MRI of the brain including volume measurement of the hippocampus, blood-oxygen level dependent imaging, and arterial spin labeling perfusion scans. On entry, patients will have CDR stage of at least 0.5 and at least one abnormal imaging biomarker.

Inclusion criteria (TBI/CTE):

* Diagnosis of Traumatic Brain Injury or Chronic Traumatic Encephalopathy
* At least 18 years of age

Exclusion Criteria:

* Macular degeneration
* Subjects with scalp rash or open wounds on the scalp (for example from treatment of squamous cell cancer)
* Advanced kidney, pulmonary, cardiac or liver failure
* Advanced terminal illness
* Any active cancer or chemotherapy
* Bone marrow disorder
* Myeloproliferative disorder
* Sickle cell disease
* Primary pulmonary hypertension
* Immunocompromising conditions and/or immunosuppressive therapies
* Any other neoplastic illness or illness characterized by neovascularity
* Subjects unable to give informed consent
* Subjects who would not be able to lay down without excessive movement in a calm environment sufficiently long enough to be able to achieve sleep
* Recent surgery or dental work within 3 months of the scheduled procedure.
* Pregnancy, women who may become pregnant or are breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-01-02 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
[Depression (MDD)] Beck Depression Inventory (BDI-II) | 6 weeks
  The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.
[Anxiety] Beck Anxiety Inventory (BAI) | 6 weeks
  The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety symptoms. Each of the 21 items asks whether the patient has experienced various anxiety symptoms in the last two weeks, and if so, how severely. Each question/answer is scored on a scale value of "0" (not at all) to "3" (severely). Higher total scores indicate more severe anxiety symptoms. The maximum total score possible is 63 points. The standard cutoff scores are: 0-7 = minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety. A reduction in score by at least 30% is considered clinically meaningful.
[Dementia] Quick Dementia Rating Scale (QDRS) | 6 weeks
  The Quick Dementia Rating Scale (QDRS) is an interview-based tool administered by study officials to participants' caregivers used to obtain observations from a consistent source. The QDRS form consists of 10 categorical questions (5 cognitive, 5 functional), each with 5 detailed options depicting the level of impairment as either 0 (normal), 0.5 (mild/inconsistent impairment), 1 (mild/consistent impairment), 2 (moderate impairment), or 3 (severe impairment). Based on the conversion table outlined in Dr. James Galvin's research (2015), total QDRS scores were converted to Clinical Dementia Rating (CDR) scale levels ranging from 0 (normal aging), 0.5 (mild cognitive impairment), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia).
[Concussion/Traumatic Brain Injury (TBI)] Brief Pain Inventory (BPI) | 6 weeks
  Self-report measure containing a composite pain score and functional interference score. The pain subscale contains 4 questions, each with answers ranging from 0 'no pain' to 10 'pain as bad as you can imagine.' Total possible score for the pain subscale is 40 points. The functional/interference subscale contains 7 questions, with each answer ranging from 0 'does not interfere' to 10 'completely interferes.' The maximum possible score for the interference subscale is 70 points. The total overall composite BPI score is out of 100 maximum points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.
[All] Global Rating of Change (GRC) | 6 weeks
  The GRC consists of a single likert-scale ranging from "-5" (very much worse) to "0" (neutral/no change) to "5" (very much better). The GRC is obtained in an interview format to assess a patient's perceived change in status following a treatment. A score that is at least 2 or greater is considered to indicate clinically significant change.

SECONDARY OUTCOMES:
[MDD & TBI] Patient Depression Questionnaire (PDQ-9) | 6 weeks
  The PDQ-9 is a 9-item, self-report questionnaire to evaluate for depressive symptoms. Each question asks the patient if they have experienced a particular depressive symptom over the past two weeks. Answers may range from "0" (not at all), "1" (several days/week), "2" (more than half of the days), and "3" (nearly every day). Maximum total score is 27 points. A higher score indicates more severe depressive symptoms. A reduction in total score by at least 30% is considered clinically meaningful.
[MDD & TBI] Patient Depression Questionnaire (PDQ-9) | 4 weeks post last day of treatment
  The PDQ-9 is a 9-item, self-report questionnaire to evaluate for depressive symptoms. Each question asks the patient if they have experienced a particular depressive symptom over the past two weeks. Answers may range from "0" (not at all), "1" (several days/week), "2" (more than half of the days), and "3" (nearly every day). Maximum total score is 27 points. A higher score indicates more severe depressive symptoms. A reduction in total score by at least 30% is considered clinically meaningful.
[MDD] Hamilton Depression Rating Scale (HAM-D) | 6 weeks
  The HAM-D is a 17-item, interview style questionnaire. A trained staff member administers this form to a patient and scores the patients' responses on a scale of "0" (symptom absent) to "4" (most severe option per symptom). A higher total score indicates a more severe level of depression. The maximum possible score is 50 points. A change in score of at least 30% is considered clinically meaningful.
[MDD] Hamilton Depression Rating Scale (HAM-D) | 4 weeks post last day of treatment
  The HAM-D is a 17-item, interview style questionnaire. A trained staff member administers this form to a patient and scores the patients' responses on a scale of "0" (symptom absent) to "4" (most severe option per symptom). A higher total score indicates a more severe level of depression. The maximum possible score is 50 points. A change in score of at least 30% is considered clinically meaningful.
[Anxiety] Hamilton Anxiety Rating Scale (HAM-A) | 6 weeks
  The HAM-A is an observer/rater scale consisting of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
[Anxiety] Hamilton Anxiety Rating Scale (HAM-A) | 4 weeks post last day of treatment
  The HAM-A is an observer/rater scale consisting of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
[Dementia] Repeatable Battery Assessment of Neuropsychological Status (RBANS) versions A-D | 6 weeks
  RBANS assesses immediate memory, visuospatial skill, language, attention, and delayed memory. Patient performance on each subscale immediate memory, language, attention, visuospatial, and delayed memory are scored relative to validated norms for same-aged peers. A change of 8+ points in the Total Scale score, 11+ points in the Immediate Memory score, 9+ points in the Language score, 4+ points on the Attention score, 14+ points is considered significant for the Visuospatial score, and 10+ points for the Delayed Memory score are considered significant.
[Dementia] Repeatable Battery Assessment of Neuropsychological Status (RBANS) versions A-D | 4 weeks post last day of treatment
  RBANS assesses immediate memory, visuospatial skill, language, attention, and delayed memory. Patient performance on each subscale immediate memory, language, attention, visuospatial, and delayed memory are scored relative to validated norms for same-aged peers. A change of 8+ points in the Total Scale score, 11+ points in the Immediate Memory score, 9+ points in the Language score, 4+ points on the Attention score, 14+ points is considered significant for the Visuospatial score, and 10+ points for the Delayed Memory score are considered significant.
[Dementia] Montreal Cognitive Assessment (MoCA) versions 7.1-7.3 | 6 weeks
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.
[Dementia] Montreal Cognitive Assessment (MoCA) versions 7.1-7.3 | 4 weeks post last day of treatment
  The MoCA evaluates frontal-executive functions (e.g., verbal abstraction and mental calculation), language (e.g., confrontation naming, phonemic fluency), orientation (e.g., person, place, date, day of the week, and time), visuospatial construction (e.g., simple figure copy), divided visual attention, and immediate and delayed memory of unstructured information. MoCA scores range from 0-30 possible points; 26 or greater is considered to reflect normal cognitive status.
[MDD] Beck Depression Inventory (BDI-II) | 4 weeks post last day of treatment
  The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.
[Anxiety] Beck Anxiety Inventory (BAI) | 4 weeks post last day of treatment
  The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety symptoms. Each of the 21 items asks whether the patient has experienced various anxiety symptoms in the last two weeks, and if so, how severely. Each question/answer is scored on a scale value of "0" (not at all) to "3" (severely). Higher total scores indicate more severe anxiety symptoms. The maximum total score possible is 63 points. The standard cutoff scores are: 0-7 = minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety. A reduction in score by at least 30% is considered clinically meaningful.
[Dementia] Quick Dementia Rating Scale (QDRS) | 4 weeks post last day of treatment
  The Quick Dementia Rating Scale (QDRS) is an interview-based tool administered by study officials to participants' caregivers used to obtain observations from a consistent source. The QDRS form consists of 10 categorical questions (5 cognitive, 5 functional), each with 5 detailed options depicting the level of impairment as either 0 (normal), 0.5 (mild/inconsistent impairment), 1 (mild/consistent impairment), 2 (moderate impairment), or 3 (severe impairment). Based on the conversion table outlined in Dr. James Galvin's research (2015), total QDRS scores were converted to Clinical Dementia Rating (CDR) scale levels ranging from 0 (normal aging), 0.5 (mild cognitive impairment), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia).
[TBI] Brief Pain Inventory (BPI) | 4 weeks post last day of treatment
  Self-report measure containing a composite pain score and functional interference score. The pain subscale contains 4 questions, each with answers ranging from 0 'no pain' to 10 'pain as bad as you can imagine.' Total possible score for the pain subscale is 40 points. The functional/interference subscale contains 7 questions, with each answer ranging from 0 'does not interfere' to 10 'completely interferes.' The maximum possible score for the interference subscale is 70 points. The total overall composite BPI score is out of 100 maximum points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.
[All] Global Rating of Change (GRC) | 4 weeks post last day of treatment
  The GRC consists of a single likert-scale ranging from "-5" (very much worse) to "0" (neutral/no change) to "5" (very much better). The GRC is obtained in an interview format to assess a patient's perceived change in status following a treatment. A score that is at least 2 or greater is considered to indicate clinically significant change.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, M.D., Principal Investigator — Neurological Associates of West Los Angeles
Locations (1):
- Neurological Associates of West Los Angele, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No
Data from this study will not be made publicly available due to ethical and privacy concerns. Anonymized data will be available upon reasonable request from any qualified investigator

REFERENCES:
- [Background] Alosco ML, Stein TD, Tripodis Y, Chua AS, Kowall NW, Huber BR, Goldstein LE, Cantu RC, Katz DI, Palmisano JN, Martin B, Cherry JD, Mahar I, Killiany RJ, McClean MD, Au R, Alvarez V, Stern RA, Mez J, McKee AC. Association of White Matter Rarefaction, Arteriolosclerosis, and Tau With Dementia in Chronic Traumatic Encephalopathy. JAMA Neurol. 2019 Nov 1;76(11):1298-1308. doi: 10.1001/jamaneurol.2019.2244. PMID 31380975
- [Background] Asken BM, Sullan MJ, DeKosky ST, Jaffee MS, Bauer RM. Research Gaps and Controversies in Chronic Traumatic Encephalopathy: A Review. JAMA Neurol. 2017 Oct 1;74(10):1255-1262. doi: 10.1001/jamaneurol.2017.2396. PMID 28975240
- [Background] Bandelow B, Michaelis S. Epidemiology of anxiety disorders in the 21st century. Dialogues Clin Neurosci. 2015 Sep;17(3):327-35. doi: 10.31887/DCNS.2015.17.3/bbandelow. PMID 26487813
- [Background] Chauhan NB. Chronic neurodegenerative consequences of traumatic brain injury. Restor Neurol Neurosci. 2014;32(2):337-65. doi: 10.3233/RNN-130354. PMID 24398724
- [Background] Cipriani A, Furukawa TA, Salanti G, Geddes JR, Higgins JP, Churchill R, Watanabe N, Nakagawa A, Omori IM, McGuire H, Tansella M, Barbui C. Comparative efficacy and acceptability of 12 new-generation antidepressants: a multiple-treatments meta-analysis. Lancet. 2009 Feb 28;373(9665):746-58. doi: 10.1016/S0140-6736(09)60046-5. PMID 19185342
- [Background] Coupe P, Manjon JV, Lanuza E, Catheline G. Lifespan Changes of the Human Brain In Alzheimer's Disease. Sci Rep. 2019 Mar 8;9(1):3998. doi: 10.1038/s41598-019-39809-8. PMID 30850617
- [Background] Edwards G 3rd, Zhao J, Dash PK, Soto C, Moreno-Gonzalez I. Traumatic Brain Injury Induces Tau Aggregation and Spreading. J Neurotrauma. 2020 Jan 1;37(1):80-92. doi: 10.1089/neu.2018.6348. Epub 2019 Aug 28. PMID 31317824
- [Background] Ferrari AJ, Charlson FJ, Norman RE, Patten SB, Freedman G, Murray CJ, Vos T, Whiteford HA. Burden of depressive disorders by country, sex, age, and year: findings from the global burden of disease study 2010. PLoS Med. 2013 Nov;10(11):e1001547. doi: 10.1371/journal.pmed.1001547. Epub 2013 Nov 5. PMID 24223526
- [Background] Galgano M, Toshkezi G, Qiu X, Russell T, Chin L, Zhao LR. Traumatic Brain Injury: Current Treatment Strategies and Future Endeavors. Cell Transplant. 2017 Jul;26(7):1118-1130. doi: 10.1177/0963689717714102. PMID 28933211
- [Background] Hamblin MR. Shining light on the head: Photobiomodulation for brain disorders. BBA Clin. 2016 Oct 1;6:113-124. doi: 10.1016/j.bbacli.2016.09.002. eCollection 2016 Dec. PMID 27752476
- [Background] Montenigro PH, Corp DT, Stein TD, Cantu RC, Stern RA. Chronic traumatic encephalopathy: historical origins and current perspective. Annu Rev Clin Psychol. 2015;11:309-30. doi: 10.1146/annurev-clinpsy-032814-112814. Epub 2015 Jan 12. PMID 25581233
- [Background] Montgomery SA, Baldwin DS, Riley A. Antidepressant medications: a review of the evidence for drug-induced sexual dysfunction. J Affect Disord. 2002 May;69(1-3):119-40. doi: 10.1016/s0165-0327(01)00313-5. PMID 12103459
- [Background] Ni H, Yang S, Siaw-Debrah F, Hu J, Wu K, He Z, Yang J, Pan S, Lin X, Ye H, Xu Z, Wang F, Jin K, Zhuge Q, Huang L. Exosomes Derived From Bone Mesenchymal Stem Cells Ameliorate Early Inflammatory Responses Following Traumatic Brain Injury. Front Neurosci. 2019 Jan 24;13:14. doi: 10.3389/fnins.2019.00014. eCollection 2019. PMID 30733666
- [Background] Rojas JC, Gonzalez-Lima F. Neurological and psychological applications of transcranial lasers and LEDs. Biochem Pharmacol. 2013 Aug 15;86(4):447-57. doi: 10.1016/j.bcp.2013.06.012. Epub 2013 Jun 24. PMID 23806754
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Schneider JA. Multiple Pathologic Pathways to Dementia in Football Players With Chronic Traumatic Encephalopathy. JAMA Neurol. 2019 Nov 1;76(11):1283-1284. doi: 10.1001/jamaneurol.2019.1089. No abstract available. PMID 31380933
- [Background] Takahata K, Kimura Y, Sahara N, Koga S, Shimada H, Ichise M, Saito F, Moriguchi S, Kitamura S, Kubota M, Umeda S, Niwa F, Mizushima J, Morimoto Y, Funayama M, Tabuchi H, Bieniek KF, Kawamura K, Zhang MR, Dickson DW, Mimura M, Kato M, Suhara T, Higuchi M. PET-detectable tau pathology correlates with long-term neuropsychiatric outcomes in patients with traumatic brain injury. Brain. 2019 Oct 1;142(10):3265-3279. doi: 10.1093/brain/awz238. PMID 31504227
- [Background] Vella MA, Crandall ML, Patel MB. Acute Management of Traumatic Brain Injury. Surg Clin North Am. 2017 Oct;97(5):1015-1030. doi: 10.1016/j.suc.2017.06.003. PMID 28958355
- [Background] Willis MD, Robertson NP. Chronic traumatic encephalopathy: identifying those at risk and understanding pathogenesis. J Neurol. 2017 Jun;264(6):1298-1300. doi: 10.1007/s00415-017-8508-x. No abstract available. PMID 28516328